CLINICAL TRIAL: NCT01054339
Title: A Multiple-Site, Phase 2, Safety and Efficacy Trial of a Recombinant Adeno-associated Virus Vector Expressing Alpha-1 Antitrypsin (rAAV1-CB-hAAT) in Patients With Alpha-1 Antitrypsin Deficiency
Brief Title: Safety & Efficacy Study of rAAV1-CB-hAAT for Alpha-1 Antitrypsin Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-AAT-002; 2009-014286-20 (Registry Identifier: EudraCT); R01HL069877 (NIH); R01FD003896 (FDA)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2016-07

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: Alpha-1 antitrypsin deficiency; Adeno-associated virus vector; AAV; Gene therapy; Human gene transfer
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): rAAV1-CB-hAAT at dosage level of 6 x 10e11 vg/kg
  Interventions: Drug: rAAV1-CB-hAAT
- Middle dose (Experimental): rAAV1-CB-hAAT at dosage level of 1.9 x 10e12 vg/kg
  Interventions: Drug: rAAV1-CB-hAAT
- High dose (Experimental): rAAV1-CB-hAAT at dosage level of 6 x 10e12 vg/kg
  Interventions: Drug: rAAV1-CB-hAAT

INTERVENTIONS:
Drug: rAAV1-CB-hAAT — Recombinant adeno-associated virus vector expressing human alpha-1 antitrypsin

SUMMARY:
Assessment of the safety and efficacy of intramuscular (IM) administration of a recombinant adenoassociated virus (rAAV) alpha-1 antitrypsin (AAT) vector (rAAV1-CB-hAAT) in AAT-deficient adults at three dosage levels [6.0 × 10e11, 1.9 × 10e12 and 6.0 × 10e12 vector genome particles (vg) per kg body weight].

Funding Sources - The FDA Office of Orphan Products Development and NIH National Heart, Lung, and Blood Institute

DETAILED DESCRIPTION:
The study is a non-randomized, open-label, multi-center, sequential, three-arm, Phase 2 clinical trial evaluating the safety and efficacy of administration of a rAAV1-CB-hAAT vector administered by IM injection. Each participant will receive rAAV1-CB-hAAT on a single occasion. Three groups of three subjects each will receive rAAV1-CB-hAAT at dosage levels of 6 x 10e11 vg/kg, 1.9 x 10e12 vg/kg or 6 x 10e12 vg/kg by IM injection. Subjects in group 1 will receive a total of 10 IM injections distributed across a single muscle site, subjects in group 2 will receive a total of 32 IM injections distributed across three muscle sites, and subjects in group 3 will receive 100 IM injections distributed across 10 muscle sites. Each injection will be given in a volume of 1.35 mL, at the appropriate vector concentration to achieve the desired total vector dose.

The three groups were enrolled sequentially, with review of safety data by a Data and Safety Monitoring Board before enrollment of each higher dosage level group.

Safety was monitored by evaluation of adverse events, hematology and clinical chemistry parameters, histological examination of muscle biopsies, and measurement of serum antibodies to AAT. Efficacy was measured by evaluation of serum concentrations of M-specific AAT and total AAT, and serum AAT phenotype determined on isoelectric focusing gels. Additional information collected included presence of the vector in blood or semen, changes in serum anti-AAV antibody titers, and changes in T cell responses to AAV and AAT.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of AAT-deficiency, as defined by a serum AAT level of less than 11 µM and a phenotype or genotype either homozygous for PI*Z or compound heterozygous consisting of PI*Z and another allele known to be associated with disease
2. Be at least 18 and not more than 75 years of age
3. Have a forced expiratory volume at one second (FEV1) >25% of predicted value (post bronchodilator)
4. Weigh ≤ 90 kg
5. Not receiving AAT augmentation therapy currently or with the past 3 months, and not planning to begin such therapy for at least 12 months after administration of rAAV1-CB-hAAT
6. Be willing to discontinue aspirin, aspirin-containing products, and other drugs that may alter platelet function, 7 days prior to dosing, resuming no earlier than 24 hours after the dose has been administered
7. Have acceptable laboratory parameters:

   * Hemoglobin ≥ 11.2 g/dL for females, ≥ 12.8 g/dL for males,
   * White blood cell count 3,300 - 12,000 cells/mm3,
   * Platelet count 125,000 - 550,000/mm3,
   * Serum creatine kinase (CK) ≤ 3 times upper normal range for study laboratory,
   * Alanine aminotransferase (ALT) ≤ 2 times upper normal range for study laboratory,
   * Serum bilirubin ≤ 1.5 times upper normal range for study laboratory,
   * Serum creatinine within normal range for study laboratory,
   * Prothrombin time (PT) ≤ 14.5 seconds and partial thromboplastin time (PTT)

     ≤ 36 seconds,
   * Normal urine dipstick (negative glucose, negative hemoglobin, and negative or trace protein),
8. For females of childbearing potential:

   * A negative pregnancy test (urine or serum) at screening and at baseline (within 2 days before administration of study agent)
   * Agreement to consistently use barrier contraception (condoms, diaphragm or cervical cap with spermicide) or another form of contraception (e.g. intrauterine device or hormonal contraception) from the screening visit until 12 months after administration of rAAV1-CB-hAAT, for sexual activity that could lead to pregnancy
9. For males of reproductive potential, agreement to consistently use barrier contraception (condoms with spermicide) for 12 months after administration of rAAV1-CB-hAAT, for sexual activity that could lead to pregnancy,
10. Provide signed informed consent before screening

Exclusion Criteria:

1. Prior receipt of any AAV gene therapy product
2. Use of anticoagulants or anti-platelet agents within 7 days prior to study agent administration
3. History of immune response to human AAT augmentation therapy as indicated by clinical history of an adverse immune response to infusion and/or decreased therapeutic effect in combination with documentation of serum anti-AAT antibodies
4. Use of acute oral or intravenous antibiotic therapy for a respiratory infection within 28 days prior to study agent administration (long-term maintenance or chronic suppressive oral antibiotics, and antibiotics for a non-respiratory indication, are allowed)
5. Use of oral or systemic corticosteroids within 28 days prior to study agent administration
6. Use of any investigational agent, or any immunosuppressive drug(s), within 3 months prior to enrollment
7. For females of childbearing potential, a positive pregnancy test at screening or baseline (within 2 days before rAAV1-CB-hAAT administration) Note: At the Cincinnati Children's Hospital Medical Center site, women of childbearing potential were not permitted to enroll in the study.
8. Females who are breast feeding
9. Have a significant abnormal EKG finding at screening and/or cardiac disease (e.g. recent myocardial infarction or CHF) within past 6 months
10. Have had pulmonary edema or a pulmonary embolism within the past 6 months
11. Have a history of immunodeficiency or other medical condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence R. Flotte, MD, Principal Investigator — University of Massachusetts Medical School, Worcester, MA; Bruce C. Trapnell, MD, Principal Investigator — Cincinnati Children's Hospital Medical Center, Cincinnati, OH; Robert A. Sandhaus, MD, PhD, Principal Investigator — National Jewish Health, Denver, CO; Noel G. McElvaney, MB, BCh, BAO, Principal Investigator — Beaumont Hospital, Dublin, Ireland
Locations (4):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Background] Brantly ML, Chulay JD, Wang L, Mueller C, Humphries M, Spencer LT, Rouhani F, Conlon TJ, Calcedo R, Betts MR, Spencer C, Byrne BJ, Wilson JM, Flotte TR. Sustained transgene expression despite T lymphocyte responses in a clinical trial of rAAV1-AAT gene therapy. Proc Natl Acad Sci U S A. 2009 Sep 22;106(38):16363-8. doi: 10.1073/pnas.0904514106. Epub 2009 Aug 12. PMID 19706466
- [Result] Flotte TR, Trapnell BC, Humphries M, Carey B, Calcedo R, Rouhani F, Campbell-Thompson M, Yachnis AT, Sandhaus RA, McElvaney NG, Mueller C, Messina LM, Wilson JM, Brantly M, Knop DR, Ye GJ, Chulay JD. Phase 2 clinical trial of a recombinant adeno-associated viral vector expressing alpha1-antitrypsin: interim results. Hum Gene Ther. 2011 Oct;22(10):1239-47. doi: 10.1089/hum.2011.053. Epub 2011 Aug 24. PMID 21609134
- [Result] Mueller C, Chulay JD, Trapnell BC, Humphries M, Carey B, Sandhaus RA, McElvaney NG, Messina L, Tang Q, Rouhani FN, Campbell-Thompson M, Fu AD, Yachnis A, Knop DR, Ye GJ, Brantly M, Calcedo R, Somanathan S, Richman LP, Vonderheide RH, Hulme MA, Brusko TM, Wilson JM, Flotte TR. Human Treg responses allow sustained recombinant adeno-associated virus-mediated transgene expression. J Clin Invest. 2013 Dec;123(12):5310-8. doi: 10.1172/JCI70314. Epub 2013 Nov 15. PMID 24231351
- See also: Applied Genetic Technologies Corporation — http://agtc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two clinical trial sites (University of Massachusetts Medical Center and Cincinnati Children's Hospital Medical Center).
Groups:
- Low Dose: rAAV1-CB-hAAT at dosage level of 6 x 10e11 vg/kg administered as 10 IM injections distributed across a single muscle site
- Middle Dose: rAAV1-CB-hAAT at dosage level of 1.9 x 10e12 vg/kg administered as 32 IM injections distributed across three muscle sites
- High Dose: rAAV1-CB-hAAT at dosage level of 6 x 10e12 vg/kg administered as 100 IM injections distributed across 10 muscle sites
Period: Overall Study
Arm/Group | Low Dose | Middle Dose | High Dose
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Middle Dose | High Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 8
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (26.4) | 48.7 (9.3) | 54.3 (3.5) | 51.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 0 | 1 | 1 | 2
Alpha-1 antitrypsin phenotype [Number; unit: participants] — Alpha-1 antitrypsin phenotype determined by isoelectric focusing gel electrophoresis
  participants
    ZZ | 2 | 3 | 3 | 8
    SZ | 1 | 0 | 0 | 1
Serum total alpha-1 antitrypsin concentration [Mean (Standard Deviation); unit: microMolar] — Average of values at screening and baseline visits. Includes 1 phenotype SZ subject in low dose group.
  microMolar | 6.56 (2.00) | 3.54 (0.12) | 3.45 (0.25) | 4.31 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 3 or 4 Adverse Events
Time Frame: During 1 year after study agent administration
Population: Analysis based on all subjects enrolled in study.
Measure: Number; unit: participants
Groups:
- Middle Dose: rAAV1-CB-hAAT at dosage level of 1.9 x 10e12 vg/kg administered as a total of 32 IM injections distributed across three muscle sites
- High Dose: rAAV1-CB-hAAT at dosage level of 6 x 10e12 vg/kg administered as100 IM injections distributed across 10 muscle sites
Arm/Group | Low Dose | Middle Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 1

2. Secondary Outcome: Changes in Serum M-specific Alpha-1 Antitrypsin Concentration
Description: Results are the mean ± SD for pre-treatment (Screening and Baseline) and Months 6-12 values and mean ± SE for the difference between the pre-treatment and months 6-12 means for 2 subjects in the low dose group and 3 subjects in each of the other two groups. The monoclonal antibody used to determine serum M-specific AAT concentrations has very little cross-reactivity with Z type AAT but cross-reacts strongly with S type AAT, causing results for this assay to be spuriously high for subject 303 in the low dose group.
Time Frame: During months 6-12 after study agent adminsitration
Population: One subject in low dose group had AAT phenotype SZ, which made measurement of M-specific serum alpha-1 antitrypsin concentration invalid.
Measure: Mean (Standard Error); unit: nanomolar
Arm/Group | Low Dose | Middle Dose | High Dose
Number analyzed (Participants) | 2 | 3 | 3
nanomolar | 31.5 (7.56) | 71.8 (22.73) | 239.2 (27.57)

3. Secondary Outcome: Changes in Serum Total Alpha-1 Antitrypsin Concentrations
Description: Results are the mean ± SD for pre-treatment (Screening and Baseline) and Months 6-12 data and mean ± SE for the difference between the pre-treatment and months 6-12 means for 3 subjects per group.
Time Frame: During months 6-12 after study agent adminstration
Population: Analysis based on all subjects enrolled in study.
Measure: Mean (Standard Error); unit: micromolar
Arm/Group | Low Dose | Middle Dose | High Dose
Number analyzed (Participants) | 3 | 3 | 3
micromolar | 0.33 (1.14) | 0.16 (0.10) | 0.19 (0.16)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Low Dose | Middle Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=3) | Middle Dose (N=3) | High Dose (N=3)
diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — A 51 y/o man received high dose of study drug on 5 Oct 2010, diverticulitis diagnosed on 14 Mar 2011, admitted to hospital, treated with antibiotics and symptoms resolved. The adverse event was considered not related to study agent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=3) | Middle Dose (N=3) | High Dose (N=3)
Injection site discomfort (General disorders) | 2 (2) | 2 (2) | 2 (2) — Because of small sample size, adverse events are listed only for (1) those considered possibly, probably or definitely related to study agent or study agent administration procedures, or (2) that occurred in more than 1 subject in the study.
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) — One other subject in the low dose group and one other subject in the mid dose group had blood CPK increase that was not considered an adverse event.
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ecchymosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Influenza-like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site atrophy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Post-procedural discomfort (General disorders) | 2 (2) | 1 (1) | 1 (1)
Lymphadenopath (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Joint sprain
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive pulmonary diseases (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Postmastectomy lymphedema syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site hemorrhage (General disorders) | 1 (1) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural edema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study results based on small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less